CLINICAL TRIAL: NCT04588805
Title: Incidence Rate of Perioperiative Venous Thromboembolism(VTE) in Colorectal Cancer Patients : a Multicenter Prospective Observational Cohort Study
Brief Title: Incidence Rate of Perioperiative VTE in Colorectal Cancer Patients : a Multicenter Prospective Observational Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Professor, Beijing Friendship Hospital
Other Study IDs: BeijingFH ZZhang
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Incidence Rate of Perioperiative Venous Thromboembolism(VTE) in Colorectal Cancer Patients
Keywords: Venous Thromboembolism; Colorectal Cancer
MeSH Terms: conditions — Venous Thromboembolism; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal Cancer Patients

SUMMARY:
This is a multi-centered, prospective, observational study aimed at observing the Incidence Rate of Perioperiative VTE in Colorectal Cancer Patients

ELIGIBILITY:
Inclusion Criteria:

* Patients in colorectal surgery ward Clinical diagnosis of colorectal cancer Prepare for radical colorectal surgery.

Exclusion Criteria:

* Patients prepare for emergency surgery Clinical diagnosis of benign colorectal disease Patients who have joined other clinic studys

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colorectal cancer patients prepare for radical colorectal surgery in colorectal surgery wards
Sampling Method: Non-Probability Sample
Enrollment: 1217 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
ncidence Rate of Perioperiative VTE | 1 month

REFERENCES:
- [Derived] Wei Q, Wang Y, An YB, Yang ZY, Liu YS, Zhang X, Gu ZC, Yao HW; CRC-VTE investigators. Rationale and design of a prospective, multicenter, cohort study on the evaluation of postoperative Venous ThromboEmbolism incidence in patients with ColoRectal Cancer (CRC-VTE trial). Transl Cancer Res. 2022 May;11(5):1406-1412. doi: 10.21037/tcr-21-1860. PMID 35706792